CLINICAL TRIAL: NCT01119443
Title: A Multiple Dose Study With Increasing Dose for Pramipexole Extended Release (ER) Tablet (0.375 mg q.d. to 1.5 mg q.d.) in Two-way Cross-over Comparison to Investigate the Bioequivalence of 1.5 mg ER x 1 Tablet q.d. Versus 0.375 mg ER x 4 Tablets q.d. Under Fasted and Fed Conditions in Japanese Healthy Male Volunteers
Brief Title: Bioequivalence of Pramipexole Extended Release (PPX ER) 1.5mg x 1 Tablet Once Daily (q.d.) vs. PPX ER 0.375mg x 4 Tablets Under Fasted and Fed Conditions in Japanese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 248.677
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Healthy

ARMS (2):
- Treatment sequence A (Other): V4: PPX ER 1.5mg x 1 fed, V5: PPX ER 0.375mg x 4 fed, V6:: PPX ER 1.5mg x 1 fasted, V5: PPX ER 0.375mg x 4 fasted
  Interventions: Drug: PPX ER
- Treatment sequence B (Other): V4: PPX ER 0.375mg x 4 fed, V5: PPX ER 1.5mg x 1 fed, V6:: PPX ER 0.375mg x 4 fasted, V5: PPX ER 1.5mg x 1 fasted
  Interventions: Drug: PPX ER

INTERVENTIONS:
Drug: PPX ER — PPX ER 0.375mg - 1.5mg for 32 days totally
  Arms: Treatment sequence A
Drug: PPX ER — PPX ER 0.375mg - 1.5mg for 32 days totally
  Arms: Treatment sequence B

SUMMARY:
Bioequivalence between PPX ER 1.5 mg x 1 tablet q.d. and 0.375 mg PPX ER x 4 tablets q.d. under fasted and fed conditions Food effect of 1.5 mg ER x 1 tablet q.d.

ELIGIBILITY:
Inclusion criteria:

* Japanese healthy male
* 20 to 40 years of age
* body mass index (BMI) between 17.6 and 26.4 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters)

Exclusion criteria:

1. Any clinical relevance findings of the medical examination as follows

   1. Blood pressure (systolic blood pressure is lower than 110 mmHg and diastolic blood pressure is lower than 60 mmHg at the screening in either a supine or a sitting position),
   2. pulse rate,
   3. electrocardiogram [ECG]
   4. laboratory test parameters) of clinical relevance
2. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of orthostatic hypotension, fainting spells or blackouts
5. Chronic or acute infections

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 248.677.001 Boehringer Ingelheim Investigational Site, Sumida-ku, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: 1.5 mg x 1 tablet once daily (q.d.) fed -> 0.375 mg x 4 tablets q.d. fed -> 1.5 mg x 1 tablet q.d. fasted -> 0.375 mg x 4 tablets q.d. fasted
- Treatment Sequence B: 0.375 mg x 4 tablets q.d. fed -> 1.5 mg x 1 tablet q.d. fed -> 0.375 mg x 4 tablets q.d. fasted -> 1.5 mg x 1 tablet q.d. fasted
Period: Up-titration Period (10 Days)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Crossover Period 1 (5 Days)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 14
Completed | 14 | 13
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Crossover Period 2 (5 Days)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Crossover Period 3 (5 Days)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Crossover Period 4 (5 Days)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: Down-titration Period (1 Day)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0
Period: End of Study (All Patients)
Arm/Group | Treatment Sequence A | Treatment Sequence B
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Sequence A: 1.5 mg x 1 tablet q.d. fed -> 0.375 mg x 4 tablets q.d. fed -> 1.5 mg x 1 tablet q.d. fasted -> 0.375 mg x 4 tablets q.d. fasted
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.8) | 29.1 (5.4) | 29.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: AUCτ,ss (Fed Conditions)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: Serial pharmacokinetic blood samples collected before drug administration, 1, 2, 2.5, 3, 4, 6, 8, 10, 12, and 23.833 hours after drug administration
Population: One subject who discontinued the study on Day 1 of Visit 4 (the first day of the first crossover period) was excluded from Pharmacokinetic data set
Measure: Geometric Mean (Standard Deviation); unit: ng·h/mL
Groups:
- Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed: Pramipexole ER 1.5 mg x 1 tablet once a day (q.d.) under fed conditions
- Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed: Pramipexole ER 0.375 mg x 4 tablets once a day (q.d.) under fed conditions
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
ng·h/mL | 33.7 (5.89) | 32.3 (5.89)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — Bioequivalence between pramipexole ER 1.5 mg x 1 tablet q.d. and pramipexole ER 0.375 mg x 4 tablets q.d. in fed condition; ANOVA; Test/Reference Ratio of the mean x 100 = 104.2, 90% CI 2-sided [98.3 to 110.3] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: Cmax,ss (Fed Conditions)
Description: maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
ng/mL | 2.24 (0.290) | 2.13 (0.255)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 104.8, 90% CI [100.1 to 109.8] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Secondary Outcome: Cτ,ss (Fed Conditions)
Description: Concentration of the analyte in plasma at time τ at steady state
Time Frame: pharmacokinetic blood samples collected at τ (23.833 hours) after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
ng/mL | 0.711 (0.184) | 0.656 (0.217)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 108.31, 90% CI 2-sided [95.634 to 122.676] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

4. Secondary Outcome: Cmin,ss (Fed Conditions)
Description: Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
ng/mL | 0.676 (0.195) | 0.633 (0.218)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 106.85, 90% CI 2-sided [93.189 to 122.251] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

5. Secondary Outcome: Tmax,ss (Fed Conditions)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
hour | 5.67 [2.00 to 10.00] | 5.76 [2.00 to 10.00]
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 98.426, 90% CI 2-sided [84.276 to 112.58] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

6. Secondary Outcome: λz,ss (Fed Conditions)
Description: Terminal rate constant of the analyte in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: per hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
per hour | 0.0609 (0.0170) | 0.0640 (0.0169)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 95.11, 90% CI 2-sided [82.461 to 109.698] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

7. Secondary Outcome: t1/2,ss (Fed Conditions)
Description: Terminal half-life of the analyte in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
hour | 11.4 (5.02) | 10.8 (6.01)

8. Secondary Outcome: MRTpo,ss (Fed Conditions)
Description: Mean residence time of the analyte in the body at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed
Number analyzed (Participants) | 27 | 27
hour | 19.1 (6.08) | 18.4 (7.60)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fed vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 104.07, 90% CI 2-sided [91.585 to 118.263] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

9. Primary Outcome: AUCτ,ss (Fasted Conditions)
Description: Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted: Pramipexole ER 1.5 mg x 1 tablet once a day (q.d.) under fasted conditions
- Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted: Pramipexole ER 0.375 mg x 4 tablets once a day (q.d.) under fasted conditions
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
ng/mL | 31.4 (7.37) | 33.6 (5.80)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — Bioequivalence between pramipexole ER 1.5 mg x 1 tablet q.d. and pramipexole ER 0.375 mg x 4 tablets q.d. in fasted condition; ANOVA; Test/Reference Ratio of the mean x 100 = 93.6, 90% CI [86.9 to 100.8] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

10. Primary Outcome: Cmax,ss (Fasted Conditions)
Description: maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
ng/mL | 2.13 (0.359) | 2.12 (0.305)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 100.2, 90% CI 2-sided [94.0 to 106.7] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

11. Secondary Outcome: Cτ,ss (Fasted Conditions)
Description: Concentration of the analyte in plasma at time τ at steady state
Time Frame: pharmacokinetic blood samples collected at τ (23.833 hours) after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
ng/mL | 0.654 (0.342) | 0.757 (0.283)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 86.57, 90% CI 2-sided [73.583 to 101.854] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

12. Secondary Outcome: Cmin,ss (Fasted Conditions)
Description: Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
ng/mL | 0.654 (0.342) | 0.757 (0.283)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 86.57, 90% CI 2-sided [73.583 to 101.854] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

13. Secondary Outcome: Tmax,ss (Fasted Conditions)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Full Range); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
hour | 4.24 [2.00 to 8.00] | 4.28 [2.50 to 8.00]
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 99.069, 90% CI 2-sided [80.688 to 117.45] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

14. Secondary Outcome: λz,ss (Fasted Conditions)
Description: Terminal rate constant of the analyte in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: /hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
/hour | 0.0520 (0.0275) | 0.0474 (0.0239)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 109.48, 90% CI 2-sided [89.571 to 133.811] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

15. Secondary Outcome: t1/2,ss (Fasted Conditions)
Description: Terminal half-life of the analyte in plasma at steady state
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
hour | 13.3 (9.82) | 14.6 (10.8)

16. Secondary Outcome: MRTpo,ss (Fasted Conditions)
Description: Mean residence time of the analyte in the body at steady state after oral administration
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted | Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted
Number analyzed (Participants) | 27 | 27
hour | 21.2 (13.1) | 22.9 (13.7)
Statistical Analysis 1: Comparison: Pramipexole ER 1.5 mg x 1 Tablet q.d. in Fasted vs Pramipexole ER 0.375 mg x 4 Tablets q.d. in Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 9, analysis 1]; ANOVA; Test/Reference Ratio of the mean x 100 = 92.63, 90% CI 2-sided [77.871 to 110.185] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

ADVERSE EVENTS:
Time Frame: 32 days
Groups:
- Up-titration: Up-titration to 0.75mg (10 days)
- 1.5 mg q.d. Fed: 1.5 mg x 1 tablet q.d. or 0.375 mg x 4 tablets q.d. in fed condition (10days in crossover)
- 1.5 mg q.d. Fast: 1.5 mg x 1 tablet q.d. or 0.375 mg x 4 tablets q.d. in fast condition (10 days in crossover)
Arm/Group | Up-titration | 1.5 mg q.d. Fed | 1.5 mg q.d. Fast
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 5/28 | 5/28 | 0/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Up-titration (N=28) | 1.5 mg q.d. Fed (N=28) | 1.5 mg q.d. Fast (N=27)
Somnolence (Nervous system disorders) | 4 | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.